CLINICAL TRIAL: NCT05349955
Title: Effects and Safety of GUideline Algorithm Based Intervention on CaRdiovascular and Renal Outcomes in Elderly Diabetic Patients With High Cardiovascular Risk in the Community- A Cluster Randomized Controlled Trial (GUARD-Community Study)
Brief Title: Effects and Safety of Diabetic GUideline Algorithm Implementation Performed by Primary Care Physicians in the Community
Acronym: GUARD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Xiaoying Li, Chief of Endocrinology Department, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZSE 20220401
Record Dates: First submitted 2022-04-16; First posted 2022-04-27 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes; Cardiovascular Complication; Diabetic Kidney Disease
Keywords: Diabetes implementation study; Diabetes guideline algorithm; Cardiovascular disease; Chronic kidney disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies; Cardiovascular Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Guideline based comprehensive management on the diabetic patients. In brief, SGLT2i or GLP-1RA will be used in priority in elderly diabetic patients with very high/high CV risk, and blood pressure controlled under 130/80mmHg， LDL-c<1.8mmol/L in the very high-risk patients or <2.6mmol/L in the high risk patients according to ESC/EASD guidelines.
Who Masked: Outcomes Assessor
Masking Description: Outcome Assessment Committee members will be blinded to outcome assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensive guideline algorithm implementation (Experimental): SGLT2i or GLP-1RA recommended in priority in subjects at very high/high CV risk. The targets of intervention will be achieved at HbA1C <7%, blood pressure <130/80mmHg， LDL-c<1.8mmol/L at very high CV risk or <2.6mmol/L at high CV risk patients, antiplatelet as secondary prevention of ASCVD.
  Interventions: Other: Intensive guideline algorithm implementation
- Conventional guideline algorithm implementation (Active Comparator): Treatment based on the current approaches implemented by local physicians(primary care physicians). Guideline based education and consults will be conducted to primary care physicians.
  Interventions: Other: Conventional guideline algorithm implementation

INTERVENTIONS:
Other: Intensive guideline algorithm implementation — Diabetes guideline pharmacological algorithm will be implemented by primary care physicians in community. In brief, SGLT2i or GLP-1RA will be recommended to control blood glucose in priority when subjects at very high/high CV risk and meet the target HbA1C<7%, control blood pressure <130/80mmHg， LDL-c<1.8mmol/L at very high CV risk patients or <2.6mmol/L at high CV risk patients, and antiplatelet as secondary prevention of ASCVD.
  Arms: Intensive guideline algorithm implementation
Other: Conventional guideline algorithm implementation — The guideline intervention is based the guidance which the local physicians followed through self learning and education. The management of diabetes paitients will be decided by local physicians.
  Arms: Conventional guideline algorithm implementation

SUMMARY:
The Effects and Safety of Diabetic GUideline Algorithm Implementation in the Community (GUARD-Community) study is a 2-arm, cluster-randomized control trial to evaluate the effect and safety of guideline algorithm intervention performed by primary care physicians on cardiovascular and renal outcomes in elderly patients with high risk in community.

DETAILED DESCRIPTION:
Diabetes is an important public health concern. Elderly diabetic patients are characterized by a long duration and complications, including chronic kidney disease and/or cardiovascular disease. In the past 30 years, the guidelines of CDS, EASD or ADA have been frequently updated. The latest guideline on pharmacological algorithm recommend that patients with cardiovascular, renal disease or very high/high CV risk patients should be treated with anti-diabetic drugs presenting target organ protection, including SGLT2i and GLP1RA. And the guideline recommend comprehensive control of the cardiovascular risk factors, such as hypertension and dyslipidemia.

This GUARD-Community study is a community based cluster-randomized controlled trial and will enroll 5600 or more participants in more than 120 clusters aged ≥ 65 years with T2DM and complicated with high/very high cardiovascular risk factors . The trial will evaluate the the effects and safety of intensive "Guideline" algorithm implementation on CVD and renal outcomes. The primary hypothesis is that guideline algorithm intervention implemented by primary care physicians will significantly reduce the risk of 4-point MACE (comprised of cardiovascular death, nonfatal myocardial infarction, nonfatal stroke or hospitalization of heart failure) rates. In Phase 1 study, the control of blood sugar, blood pressure and lipids will be evaluated at 18 months after intervention. In Phase 2 study, the CVD and renal outcomes will be evaluated at 3 years. The study will last for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* ①Males or females aged 65 and above (≥65) receive treatment from the local community health service center;
* ②Diagnosed type 2 diabetes (ADA criteria):
* A. Typical symptoms of diabetes + random blood sugar ≥ 11.1mmol/L;
* B. Fasting blood glucose (FPG) ≥ 7.0mmol/L (fasting blood glucose is defined as no caloric intake within 8 hours);
* C. Oral glucose tolerance test 2h blood glucose (OGTT) ≥ 11.1mmol/L (2h after meal);
* D. have been treated with antidiabetic drugs;
* Each blood sugar test must be repeated to confirm the diagnosis;
* ③Complicated with chronic kidney disease and/or very high/high risk of cardiovascular disease, meet any one of the following:
* A. ASCVD, including coronary heart disease, cerebral infarction, peripheral vascular disease;
* B. Or target organ damage (albuminuria, renal impairment with eGFR ≥ 30 ml/min/1.73m2, left ventricular hypertrophy or retinopathy);
* C. ≥ 3 major risk factors (age ≥ 65 years old, hypertension, dyslipidemia, smoking, obesity );
* D. Diabetes duration ≥ 10 years, with any one traditional cardiovascular risk factor such as advanced age, obesity, smoking, sedentary, family history of cardiovascular disease, hypertension, abnormal lipid metabolism.

Exclusion Criteria:

* ①Pregnant women or women planning to become pregnant;
* ②eGFR<30 mL/min/1.73m2 (CKD-EPI formula);
* ③Patient cannot be followed up for 36 months (due to health condition or migration);
* ④Unwilling or unable to sign the informed consent;
* ⑤Type 1 diabetes;

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5600 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome of Phase 1: Comprehensive management effect of various cardiovascular risk factors in T2D，meeting control targets for a combination of A1c, BP, LDL-C. | 18 months since randomization
  The proportion of participants with HbA1C<7.0%, blood pressure< 130/80 mm Hg，LDL-c<1.8mmol/L at very high CV risk or <2.6mmol/L at high CV risk.
Primary Outcome of Phase 2: Composite of 3P MACE and hospitalization for heart failure. | 3 years since randomization
  Time to occurrence of cardiovascular and cerebrovascular death, non-fatal myocardial infarction, non-fatal Stroke, hospitalization for heart failure.

SECONDARY OUTCOMES:
Secondary Outcome of Phase 1: Glycemic control rate | 18 months since randomization
  The proportion of participants with tight glucose control, targeting HbA1c <7.0%
Secondary Outcome of Phase 1: Mean HbA1C changes | 18 months since randomization
  Mean HbA1C changes of participants
Secondary Outcome of Phase 1: Mean systolic and diastolic pressure changes | 18 months since randomization
  Mean systolic and diastolic pressure changes of participants
Secondary Outcome of Phase 1: Mean LDL-c changes | 18 months since randomization
  Mean LDL-c changes of participants
Secondary Outcome of Phase 1: Adherence to guideline algorithm medication recommendation rate | 18 months since randomization
  Use electronic medical recorded prescription and questionnaires to assess the proportion of participants who adhere to guideline recommended medication
Secondary Outcome of Phase 2: Incident or worsening nephropathy | 3 years since randomization
  Time to composite of incident macroalbuminuria (UACR >300 mg/g), a sustained decline in eGFR (decrease in the eGFR of 30% or more to a value of less than 60 when baseline ≥60ml per minute per 1.73 m2, decrease in the eGFR of 50% or more when baseline <60ml per minute per 1.73 m2)from baseline, or chronic renal replacement therapy, or renal death.
Secondary Outcome of Phase 2: Cardiorenal composite endpoint | 3 years since randomization
  Time to eGFR (CKD-EPI formula) decrease, renal replacement therapy, renal or cardiovascular death
Secondary Outcome of Phase 2: 3P MACE | 3 years since randomization
  Time to events occurence: cardiovascular death, non-fatal myocardial infarction, non-fatal stroke
Secondary Outcome of Phase 2: New onset of macroalbuminuria. | 3 years since randomization
  Time to UACR>300mg/g
Secondary Outcome of Phase 2: Changes of myocardial ischemia in electrocardiogram (ECG) | 3 years since randomization
  Participants number of ECG ischemia demonstration occurence: ST-T segment depression more than 0.1mv in two adjacent leads of ECG compared with baseline, poor R wave progression.
Secondary Outcome of Phase 2: New onset of albuminuria | 3 years since randomization
  Time to UACR increase from <30mg/g to ≥30mg/g
Secondary Outcome of Phase 2: Albuminuria progression | 3 years since randomization
  Time to albuminuria progression: UACR increased by ≥30% and grade progression (ie, from normal to micro or macro, or from micro to macro)
Secondary Outcome of Phase 2: Albuminuria regression | 3 years since randomization
  Time to albuminuria regression: UACR grade regression(ie, from macro to micro or normal, or from micro to normal), and the UACR value decreases by more than or equal to 30%
Secondary Outcome of Phase 2: Changes in the ratio of patients with normal or abnormal urine protein at the end of the study | 3 years since randomization
  Rate change of normal or abnormal UACR. Normal means UACR<30mg/g. Abnormal means UACR≥30mg/g
Secondary Outcome of Phase 2: Slope of eGFR decline | 3 years since randomization
  Decrease of the eGFR over time
Secondary Outcome of Phase 2: Retinopathy changes | 3 years since randomization
  Occurrence or regression of retinopathy(ETDRS-DRSS)
Secondary Outcome of Phase 2: Body weight change | 3 years since randomization
  Absolute weight change and the percentage change of body weight
Secondary Outcome of Phase 2: Changes of fatty liver prevalence | 3 years since randomization
  Rate change of fatty liver.
Secondary Outcome of Phase 2: Changes in beta-cell function | 3 years since randomization
  Absolute change assessed by HOMA2-%β method
Secondary Outcome of Phase 2: Changes in cognitive function | 3 years since randomization
  Improvement or progression of cognitive function: The Mini-CogTM scale
Secondary Outcome of Phase 2: The FRAIL scale | 3 years since randomization
  Changes of the simple frailty questionnaire score
Secondary Outcome of Phase 2: All-cause death | 3 years since randomization
  Time to the death due to any cause

OTHER OUTCOMES:
Health Economics Indicators | 3 years since randomization
  Cost-effectiveness analysis： quantification of Incremental Cost Ratio Life Cycle (ICER) and Quality Adjusted Years (QALYs)
Changes in cardiovascular risk indicators | 3 years since randomization
  Framingham score
Serology and urine testing | 3 years since randomization
  Biomarkers associated with diagnosis or prognosis: using "omics" screening.
Genomics testing | 3 years since randomization
  Gene polymorphism testing for drug response or prognosis: using genome-wide association study(GWAS) screening.
The time rate of glycemic target range | 3 years since randomization
  Continous glucose monitor detection

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Li, MD, Principal Investigator — Fudan University
Locations (13):
- China (13):
  - Xiangcheng Second People's Hospital, Suzhou, Jaingsu
  - Caohu Community Healthcare Center, Suzhou, Jiangsu
  - Huangqiao Community Healthcare Center, Suzhou, Jiangsu
  - Xiangcheng People's Hospital., Suzhou, Jiangsu
  - Yuanhe Community Healthcare Center, Suzhou, Jiangsu
  - Xiangcheng Third People's Hospital, Suzhou, Jiangsu
  - Taiping Community Healthcare Center, Suzhou, Jiangsu
  - Yangchenghu People's Hospital, Suzhou, Jiangsu
  - Health Center of Xiangcheng Tourism Resort, Suzhou, Jiangsu
  - Caohu People's Hospital, Suzhou, Jiangsu
  - Dongqiao Community Healthcare Center, Suzhou, Jiangsu
  - Xiangcheng Traditional Chinese Medicine Hospital, Suzhou, Jiangsu
  - Chengyang Community Healthcare Center, Suzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No
The data will be available from the principle investigator on reasonable request.

REFERENCES:
- [Background] Gu TW, Zhu DL. [Interpretation of treatment part of national guideline for the prevention and control of diabetes in primary care (2018)]. Zhonghua Nei Ke Za Zhi. 2019 Jul 1;58(7):538-540. doi: 10.3760/cma.j.issn.0578-1426.2019.07.011. Chinese. PMID 31269573
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Gross JL, de Azevedo MJ, Silveiro SP, Canani LH, Caramori ML, Zelmanovitz T. Diabetic nephropathy: diagnosis, prevention, and treatment. Diabetes Care. 2005 Jan;28(1):164-76. doi: 10.2337/diacare.28.1.164. PMID 15616252
- [Background] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Background] Wiviott SD, Raz I, Bonaca MP, Mosenzon O, Kato ET, Cahn A, Silverman MG, Zelniker TA, Kuder JF, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Ruff CT, Gause-Nilsson IAM, Fredriksson M, Johansson PA, Langkilde AM, Sabatine MS; DECLARE-TIMI 58 Investigators. Dapagliflozin and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2019 Jan 24;380(4):347-357. doi: 10.1056/NEJMoa1812389. Epub 2018 Nov 10. PMID 30415602
- [Background] Neal B, Perkovic V, Mahaffey KW, de Zeeuw D, Fulcher G, Erondu N, Shaw W, Law G, Desai M, Matthews DR; CANVAS Program Collaborative Group. Canagliflozin and Cardiovascular and Renal Events in Type 2 Diabetes. N Engl J Med. 2017 Aug 17;377(7):644-657. doi: 10.1056/NEJMoa1611925. Epub 2017 Jun 12. PMID 28605608
- [Background] Bhatt DL, Szarek M, Steg PG, Cannon CP, Leiter LA, McGuire DK, Lewis JB, Riddle MC, Voors AA, Metra M, Lund LH, Komajda M, Testani JM, Wilcox CS, Ponikowski P, Lopes RD, Verma S, Lapuerta P, Pitt B; SOLOIST-WHF Trial Investigators. Sotagliflozin in Patients with Diabetes and Recent Worsening Heart Failure. N Engl J Med. 2021 Jan 14;384(2):117-128. doi: 10.1056/NEJMoa2030183. Epub 2020 Nov 16. PMID 33200892
- [Background] Heerspink HJL, Stefansson BV, Correa-Rotter R, Chertow GM, Greene T, Hou FF, Mann JFE, McMurray JJV, Lindberg M, Rossing P, Sjostrom CD, Toto RD, Langkilde AM, Wheeler DC; DAPA-CKD Trial Committees and Investigators. Dapagliflozin in Patients with Chronic Kidney Disease. N Engl J Med. 2020 Oct 8;383(15):1436-1446. doi: 10.1056/NEJMoa2024816. Epub 2020 Sep 24. PMID 32970396
- [Background] Perkovic V, Jardine MJ, Neal B, Bompoint S, Heerspink HJL, Charytan DM, Edwards R, Agarwal R, Bakris G, Bull S, Cannon CP, Capuano G, Chu PL, de Zeeuw D, Greene T, Levin A, Pollock C, Wheeler DC, Yavin Y, Zhang H, Zinman B, Meininger G, Brenner BM, Mahaffey KW; CREDENCE Trial Investigators. Canagliflozin and Renal Outcomes in Type 2 Diabetes and Nephropathy. N Engl J Med. 2019 Jun 13;380(24):2295-2306. doi: 10.1056/NEJMoa1811744. Epub 2019 Apr 14. PMID 30990260
- [Background] Marso SP, Daniels GH, Brown-Frandsen K, Kristensen P, Mann JF, Nauck MA, Nissen SE, Pocock S, Poulter NR, Ravn LS, Steinberg WM, Stockner M, Zinman B, Bergenstal RM, Buse JB; LEADER Steering Committee; LEADER Trial Investigators. Liraglutide and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2016 Jul 28;375(4):311-22. doi: 10.1056/NEJMoa1603827. Epub 2016 Jun 13. PMID 27295427
- [Background] Gerstein HC, Colhoun HM, Dagenais GR, Diaz R, Lakshmanan M, Pais P, Probstfield J, Riesmeyer JS, Riddle MC, Ryden L, Xavier D, Atisso CM, Dyal L, Hall S, Rao-Melacini P, Wong G, Avezum A, Basile J, Chung N, Conget I, Cushman WC, Franek E, Hancu N, Hanefeld M, Holt S, Jansky P, Keltai M, Lanas F, Leiter LA, Lopez-Jaramillo P, Cardona Munoz EG, Pirags V, Pogosova N, Raubenheimer PJ, Shaw JE, Sheu WH, Temelkova-Kurktschiev T; REWIND Investigators. Dulaglutide and cardiovascular outcomes in type 2 diabetes (REWIND): a double-blind, randomised placebo-controlled trial. Lancet. 2019 Jul 13;394(10193):121-130. doi: 10.1016/S0140-6736(19)31149-3. Epub 2019 Jun 9. PMID 31189511
- [Background] Marso SP, Bain SC, Consoli A, Eliaschewitz FG, Jodar E, Leiter LA, Lingvay I, Rosenstock J, Seufert J, Warren ML, Woo V, Hansen O, Holst AG, Pettersson J, Vilsboll T; SUSTAIN-6 Investigators. Semaglutide and Cardiovascular Outcomes in Patients with Type 2 Diabetes. N Engl J Med. 2016 Nov 10;375(19):1834-1844. doi: 10.1056/NEJMoa1607141. Epub 2016 Sep 15. PMID 27633186
- [Background] Cosentino F, Grant PJ, Aboyans V, Bailey CJ, Ceriello A, Delgado V, Federici M, Filippatos G, Grobbee DE, Hansen TB, Huikuri HV, Johansson I, Juni P, Lettino M, Marx N, Mellbin LG, Ostgren CJ, Rocca B, Roffi M, Sattar N, Seferovic PM, Sousa-Uva M, Valensi P, Wheeler DC; ESC Scientific Document Group. 2019 ESC Guidelines on diabetes, pre-diabetes, and cardiovascular diseases developed in collaboration with the EASD. Eur Heart J. 2020 Jan 7;41(2):255-323. doi: 10.1093/eurheartj/ehz486. No abstract available. PMID 31497854
- [Background] American Diabetes Association. 9. Pharmacologic Approaches to Glycemic Treatment: Standards of Medical Care in Diabetes-2021. Diabetes Care. 2021 Jan;44(Suppl 1):S111-S124. doi: 10.2337/dc21-S009. PMID 33298420
- [Background] Mosenzon O, Wiviott SD, Heerspink HJL, Dwyer JP, Cahn A, Goodrich EL, Rozenberg A, Schechter M, Yanuv I, Murphy SA, Zelniker TA, Gause-Nilsson IAM, Langkilde AM, Fredriksson M, Johansson PA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Sabatine MS, Raz I. The Effect of Dapagliflozin on Albuminuria in DECLARE-TIMI 58. Diabetes Care. 2021 Aug;44(8):1805-1815. doi: 10.2337/dc21-0076. Epub 2021 Jul 7. PMID 34233928
- [Background] Wanner C, Inzucchi SE, Lachin JM, Fitchett D, von Eynatten M, Mattheus M, Johansen OE, Woerle HJ, Broedl UC, Zinman B; EMPA-REG OUTCOME Investigators. Empagliflozin and Progression of Kidney Disease in Type 2 Diabetes. N Engl J Med. 2016 Jul 28;375(4):323-34. doi: 10.1056/NEJMoa1515920. Epub 2016 Jun 14. PMID 27299675